CLINICAL TRIAL: NCT05411640
Title: Effect of Blood Flow Restriction Training on Glycemic Control, Functional Activity and Quality of Life in Individuals With Prediabetes
Brief Title: Effect of BFR Training on Glycemic Control, Functional Activity and Quality of Life in Individuals With Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/1103
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: PreDiabetes
Keywords: Prediabetic State; Glycemic Control
MeSH Terms: conditions — Prediabetic State | interventions — Exercise; Patient Education as Topic; Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobics with Blood flow restriction (Experimental): This group will perform Aerobic exercises with Blood Flow Restriction training, patient education and dietary modifications will be given for pre diabetes
  Interventions: Other: Aerobic exercise with Blood flow restriction
- Aerobics without Blood flow restriction (Active Comparator): This group will perform Aerobic exercises without Blood Flow Restriction training, patient education and dietary modifications will be given for pre diabetes.
  Interventions: Other: Aerobic exercise without Blood flow restriction
- Education and Dietary modifications (Other): This group will only receive education and dietary modifications for Pre-diabetes.
  Interventions: Other: Patient Education and dietary modification

INTERVENTIONS:
Other: Aerobic exercise with Blood flow restriction — Experimental group will be given aerobic exercises with blood flow restriction training. For first four weeks, aerobic exercise will be performed for 25 min with 60-65 % of the maximum heart rate reserve (MHRR). During second four weeks, time of exercise will be 30 min with intensity 60-65% of the MHRR, and for third four weeks, time will be increased to 35 min and intensity will be raised up to 70-75% of the MHRR. . Arterial occlusion of 60% will be achieved by Blood Flow Restriction apparatus. Total intervention protocol for this group will be given for 12 weeks of duration 4 sessions per week with total 48 sessions.
  Arms: Aerobics with Blood flow restriction
Other: Aerobic exercise without Blood flow restriction — Active Comparator group will be given aerobic exercises. For first four weeks, aerobic exercise will be performed for 25 min with 60-65 % of the maximum heart rate reserve (MHRR). During second four weeks, time of exercise will be 30 min with intensity 60-65% of the MHRR, and for third four weeks, time will be increased to 35 min and intensity will be raised up to 70-75% of the MHRR. Total intervention protocol for this group will be given for 12 weeks of duration 4 sessions per week with total 48 sessions.
  Arms: Aerobics without Blood flow restriction
Other: Patient Education and dietary modification — Participants will individually instruct to reduce total energy intake and increase physical activity, aiming at a 5% reduction in body weight. The participants will be given pamphlets providing general information on pre diabetes and dietary modifications. Total intervention protocol for the group will be given for 12 weeks of duration 4 sessions per week with total 48 sessions.
  Arms: Education and Dietary modifications

SUMMARY:
The aim of this study is to determine the effects of blood flow restriction training on glycemic control and functional activity in participants with prediabetes. Moreover, This study determine the effects of blood flow restriction training on quality of life in participants with prediabetes

DETAILED DESCRIPTION:
In 2021, a randomized control trial had been conducted to determine the effects of two methods of resistance training with and without blood flow restriction on coagulation indices and blood glucose levels in type 2 diabetic patients. This study recruited 41 patients with type 2 diabetes were randomly divided into three groups of resistance training with and without blood flow restriction and the control group. The subjects of the resistance training group with and without flow restriction performed the training for 8 weeks with intensities of 20, 40, 60, 80% of one maximum repetition and 20 and 30% of one maximum repetition, respectively. During this period, the subjects in the control group led a normal life and did not have a regular exercise program. Coagulation parameters, hematocrit and blood glucose levels were measured before and 48 hours after the last training session. This study concluded that 8 weeks of resistance training can prevent thrombosis and sudden onset of cardiovascular disease in patients with type 2 diabetes by reducing fibrinogen levels and increasing the Prothrombin Time index. This type of exercise also plays an insulin-like role by lowering blood sugar levels.

In 2019, a randomized control trial had been conducted to determine the Proximal, Distal, and Contralateral Effects of Blood Flow Restriction Training on the Lower Extremities. This study included 26 patients, providing 16 Blood Flow Restriction and 10 control patients. Patients were excluded for cardiac, pulmonary, or hematologic disease; pregnancy; or previous surgery in the extremity. The experimental group completed a standardized 6-week course of Blood Flow Restriction training. All participants of experimental group completed the following exercises at each training session: straight-leg raise hip flexion, side-lying hip abduction, long-arc quadriceps extension, and standing hamstring curl. Strength exercises were performed on both extremities using predetermined weight, calculated as 30% of 1-repitition (rep) maximum determined 1 week prior to the initiation of training Data collected at baseline and completion included limb circumferences and strength testing. This study concluded that low-load Blood Flow Restriction training increased muscle strength and limb circumference more than high- load Blood Flow Restriction training. Both the proximal and distal muscle groups were strengthened by Blood Flow Restriction exercise. A systemic or crossover effect could be confirmed by gains in the contralateral extremity.

In 2019, a randomized control trial had been conducted to determine the effects of Low-load blood flow restriction training that induces similar morphological and mechanical Achilles' tendon adaptations as compared with high-load resistance training. This study included 55 male volunteers those were randomly allocated into the following three groups: low load- Blood Flow Restriction, high load and a non-exercising control group. The low load- Blood Flow Restriction and high load groups completed a resistance training program for 14 week, and tendon morphology, mechanical as well as material properties, and muscle cross- sectional area and isometric strength were assessed before and after the intervention. This study concluded that the adaptive change in Achilles' tendon properties following low-load resistance training with partial vascular occlusion appears comparable to that evoked by high-load resistance training.

In 2018, a randomized control trial had been conducted to determine the effects of lower body blood flow restriction training may induce remote muscle strength adaptations in an active unrestricted arm. 24 participants were recruited in this study which were divided in two groups. an experimental Blood Flow Restriction group (EXP; n = 12) or a non- Blood Flow Restriction control group (CON; n = 12) completed 7-weeks of resistance training comprising three sets of unilateral bicep curls [50% 1-repetition maximum (1-RM)], then four sets of bilateral knee extension and flexion exercises (30% 1-RM). Experimental group performed leg exercises with an applied Blood Flow Restriction (60% limb occlusion pressure). 1-RM strength was measured using bilateral leg exercises and unilateral bicep curls in both trained and untrained arms. Muscle CSA was measured via peripheral quantitative computed tomography in the dominant leg and both arms. This study concluded that Blood Flow Restriction training increased trained arm strength more than the contralateral untrained arm, and the trained arm of control.

In 2018, a randomized control trial had been conducted to determine the effects of benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. This study recruited forty-eight women with knee OA were randomized into one of the three groups: low-intensity resistance training (30% one repetition maximum 1-RM) associated (BFRT) or not (LI-RT) with partial blood flow restriction, and high-intensity resistance training (HI- RT: 80% 1-RM). Patients underwent a 12-week supervised training program and were assessed for lower-limb 1-RM, quadriceps cross-sectional area (CSA), functionality (timed stands test - TST and timed-up-and-go test - TUG), and disease-specific inventory (Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC) before (PRE) and after the protocol (POST). This study concluded that BFRT and HI-RT were similarly effective in increasing muscle strength, quadriceps muscle mass, and functionality in knee OA patients. Importantly, BFRT was also able to improve pain while inducing less joint stress, emerging as a feasible and effective therapeutic adjuvant in OA management.

In previous studies, blood flow restriction technique has been used in clinical practice to increase the muscle mass and muscle strength. Literature is limited regarding the effects of Blood Flow Restriction to treat and control pre diabetes. Moreover, there are very less evidence that studied about the effect of Blood Flow Restriction to prevent the progression to diabetes mellites in pre-diabetic participants. Therefore, current study is designed to determine the effects of blood flow restriction training on glycemic control in individuals with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Both male & female participants
* Age group between 30 to 60 years.
* Subjects clinically diagnosed with prediabetes (41-49 mmol/mol) after fasting blood sugar (110-125 mg/dl) and Hb1Ac (5.7%-6.4%) or assessed using the diabetes risk assessment tool as having high risk of developing diabetes in the next five years.
* Mean BMI for participants will be more than 22.
* Subjects able to understand simple instructions, independently or with assistance from their support person.

Exclusion Criteria:

* History of any cardiovascular problems that limited safe participation in aerobic or resistance exercise.
* Subjects who are unable to walk 30 min independently with or without a walking aid
* History of any psychological disorder.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Sugar Level | 16th week
  This measures your blood sugar after an overnight fast (not eating). A fasting blood sugar level of 99 mg/dL or lower is normal, 100 to 125 mg/dL indicates you have prediabetes, and 126 mg/dL or higher indicates you have diabetes.
Hemoglobin A1c (HbA1c) test | 16th week
  ,A hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to hemoglobin. An HbA1c test may be used to check for diabetes or prediabetes in adults. The Centers for Disease Control (CDC) recommends that adults over the age of 45 get tested to screen for diabetes and prediabetes. HbA1c results are given in percentages. Typical results for this test are Normal value of HbA1c below 5.7%, for prediabetes, HbA1c between 5.7% and 6.4%, for diabetes, HbA1c of 6.5% or higher.
Australian type 2 diabetes risk assessment tool (AUSDRISK) | 16th week
  The Australian type 2 diabetes risk assessment tool (AUSDRISK) is a short list of questions. It helps both health professionals and individuals to assess the risk of a person developing type 2 diabetes over the next 5 years. It consists of 10 questions with each question containing 2 options. Individuals who score 5 or less than 5 are at low risk. Individuals who score 6 to 11 are at intermediate risk of developing diabetes. While, Individuals who score 12 or more are at high risk of developing diabetes

SECONDARY OUTCOMES:
World Health Organization Quality of Life | 16th week
  The World Health Organization Quality of Life (WHOQOL) consists of a set of survey questions that can be used to collect data related to an individual in particular and society in general on various parameters that determine their general quality of life, their natural environment, their health, their living condition, their community and more. There are many factors that are associated while measuring the quality of life, like physical health, physiological well-being, social relationships, functional roles and subjective sense of lifestyle satisfaction
36-Item Short Form Survey | 16th week
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study. The original authors designed the SF-36 to measure health at the individual level in clinical practice and research and at the population level for health policy evaluations, and general population surveys. It has been used in thousands of research studies. The SF-36 was originally designed as a generic health measure but has also been applied to specific disease populations. Patients or individuals are asked to fill out the questionnaire (tick boxes) by themselves and then it is scored by a clinician or researcher
International Physical Activity Questionnaires | 16th week
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires. Long (5 activity domains asked independently) and short (4 generic items) versions for use by self- administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity. IPAQ can provide researchers and practitioners with an estimate of physical activity and sedentary behavior for adults aged 15-69 years, across a range of socio-economic settings
Rockport Walking Fitness Test | 16th week
  Rockport Walking Fitness Test also known as 1-mile walk test, conducted by putting a Beurer Heart Rate Monitor (PM-26) and walking in slow circles and do light stretching for 10 minutes to warm up before starting the test. Start the stopwatch and walk the entire distance of a 1 mile (1.6 km) on a treadmill. After 1 mile, turn off the stopwatch and immediately check your heart rate. Continue walking, slowly, for another 5 minutes to cool down.
Borg rating of perceived exertion | 16th week
  Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. The scale is a very simple numerical list. Participants are asked to rate their exertion on the scale during the activity, taking into consideration feelings of physical stress and fatigue, disregarding any factor such as leg pain or breathlessness but focusing on the whole feeling of exertion. This number chosen connotes the intensity of activity allowing the participant to speed up or slow down movements/activity. The scale takes
  a few seconds to complete, can be self or researcher administered on a single occasion or multiple times.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, Ph.D, Principal Investigator — Riphah International University; Muhammad Abbas, Principal Investigator — Riphah International University , QIE, Campus
Locations (1):
- Ahmad Poly care clinic, Faislabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No